CLINICAL TRIAL: NCT04023890
Title: Ventricular Electrical Synchronization by Stimulating Left and Right Bundle Branches Area in Pacing-indicated Patients
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: Bundle Branches Area Pacing
Record Dates: First submitted 2019-07-16; First posted 2019-07-18 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Cardiac Pacing; Pacing Therapy; Pacemaker

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective, single-site, non-randomized, acute feasibility clinical study. The purpose of this study is to explore the electrocardiogram (ECG) characteristics of simultaneous stimulation of right and left bundle branches area.

DETAILED DESCRIPTION:
Many pacemaker patients have cardiac conduction system disease and thus need ventricular pacing. Traditional ventricular pacing causes ventricular dyssynchrony that in turn causes cardiac contraction dysfunction. CRT pacing provides better ventricular synchronization, but not the optimal, especially in patients with narrow QRS. CRT non-response rate is at 30%. His bundle pacing utilizes naturel His bundle-Purkinjie system to provide optimal physiological pacing. But many pacing-indicated patients have abnormal His bundle-Purkinje system, thus His bundle pacing cannot provide optimal pacing in patients with abnormal cardiac conduction system. Moreover, the pacing threshold is high during His bundle pacing. More recently, left bundle branch pacing is proposed. However, LBBP will generate right bundle branch block pattern, another kind of weak ventricular synchronization. Thus, the investigators propose to excite the left and right bundle branches area simultaneously to normalize ventricular synchronization. The purpose of this study is to explore the electrocardiogram (ECG) characteristics of simultaneous stimulation of right and left bundle branches area.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 18 to 80 years old
* Subjects who are willing to provide Informed Consent
* Subjects who have pacing indications or indications for CRT, and will receive pacemaker or CRT therapy

Exclusion Criteria:

* Subjects who have contra-indications for pacing therapy or CRT
* CRT up-graded subjects
* Ventricular hypertrophy
* Subjects who have medical conditions that would limit study participation
* Subjects who are pregnant or have a plan for pregnancy during the study
* Subjects who are not willing to provide Informed Consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll subjects who have pacing indications or indications for CRT.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
QRS duration | During implant
  The primary endpoint is QRS duration during bundle branches area pacing

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohong Zhou, M.D., Study Director — Medtronic
Locations (1):
- Fuwai Hospital, Beijing, Beijing Municipality, China